CLINICAL TRIAL: NCT05148676
Title: Residual Symptoms and the Quality of Life in Individuals Recovered From COVID-19 Infection: A Survey From Pakistan
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Rubaid Azhar Dhillon, MBBS, Aga Khan University
Other Study IDs: 2021-5584-17843
Record Dates: First submitted 2021-12-07; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Pandemic; COVID-19 Respiratory Infection; COVID-19 Lower Respiratory Infection
Keywords: COVID-19; Residual Symptoms; Quality of Life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Residual Symptoms and the Quality of Life in Individuals Recovered from COVID-19 Infection: A Survey from Pakistan — An anonymous online survey was administrated in Pakistan from November 2020 to April 2021 in COVID-19 survivors. The questionnaire used the 12-Item Short Form Health Survey (SF-12) to assess mental and physical QoL. Multivariate linear regression was used to explore factors associated with mental and physical QoL scores.

SUMMARY:
There remains scarcity of literature regarding the patient's health status post-COVID-19 infection. This study analyzes the prevalence of residual symptoms and quality of life (QoL) after COVID-19.

DETAILED DESCRIPTION:
An anonymous online survey was administrated in Pakistan from November 2020 to April 2021 in COVID-19 survivors. The questionnaire used the 12-Item Short Form Health Survey (SF-12) to assess mental and physical QoL. Multivariate linear regression was used to explore factors associated with mental and physical QoL scores.

A total of 331 COVID-19 survivors participated in our survey. Around 42.0% of the cohort reported within 1-3 months of diagnosis of COVID-19. The common residual symptoms were body aches (39.9%), low mood (32.6%), and cough (30.2%). Better physical QoL was associated with being male (adjusted beta: 3.328) and having no residual symptoms (6.955). However, suffering from nausea/vomiting during initial COVID-19 infection (-4.026), being admitted to the ICU during COVID-19 infection (-9.164), and suffering from residual body aches (-5.209) and low mood (-2.959) was associated with poorer QoL. Better mental QoL was associated with being asymptomatic during initial COVID-19 infection (6.149) and post-COVID (6.685), while experiencing low mood post-COVID was associated with poorer mental QoL (-8.253 [-10.914, -5.592]).

Despite presumed "recovery" from COVID-19, patients still face a wide range of residual symptoms months after initial infection, which contributes towards poorer QoL. Healthcare professionals must remain alert to the long-lasting effects of COVID-19 infection and aim to address them appropriately to improve patients' QoL.

ELIGIBILITY:
Inclusion Criteria:

* Tested negative for COVID-19 when enrolled in the study
* COVID-19 negative for at least 6 months

Exclusion Criteria:

* Still Positive for COVID-19 tested one week ago
* COVID-19 negative for less than 6 months

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 331 individuals who responded to the online survey were included in the study. The majority were aged between 18-35 years (72.2%) and were residents of the province of Sindh (62.8%). Around half (54.1%) of the respondents were married, while 10.6% were separated or divorced. The highest level of education was reported as bachelors or lower by 45% of respondents. The common comorbidities were hypertension (9.4%), asthma (9.1%), and type 2 diabetes mellitus (7.3%).
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Residual Symptoms and the Quality of Life in Individuals Recovered from COVID-19 Infection: A Survey from Pakistan | November 2020 to April 2021
  The questionnaire used the 12-Item Short Form Health Survey (SF-12) to assess mental and physical QoL. Multivariate linear regression was used to explore factors associated with mental and physical QoL scores.

CONTACTS AND LOCATIONS:
Overall Officials: Rubaid A Dhillon, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The anonymous data collected of participants will be not shared publicly, only limited information will be displayed in the study where necessary.